CLINICAL TRIAL: NCT01183026
Title: Performance of V/Q SPECT for the Diagnosis of Pulmonary Embolism
Brief Title: V/Q SPECT for Diagnosis of Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: PENNEC, CHU de BREST
Other Study IDs: SPECT
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study was to assess diagnostic performance of V/Q SPECT for the diagnosis of pulmonary embolism by comparing V/Q SPECT results to a validated diagnostic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary embolism suspicion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary embolism suspicion
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

REFERENCES:
- [Derived] Le Duc-Pennec A, Le Roux PY, Cornily JC, Jaffrelot M, Delluc A, de Saint-Martin L, Guillo P, Le Gal G, Salaun PY, Leroyer C. Diagnostic accuracy of single-photon emission tomography ventilation/perfusion lung scan in the diagnosis of pulmonary embolism. Chest. 2012 Feb;141(2):381-387. doi: 10.1378/chest.11-0090. Epub 2011 Aug 18. PMID 21852295